CLINICAL TRIAL: NCT00773071
Title: Added-value of SPECT/CT in Patients Undergoing Lymphatic Mapping and Sentinel Lymphadenectomy (LM/SL) for Gynecological Cancers
Brief Title: Added-value of SPECT/CT in Patients Undergoing LM/SL for Gynecological Cancers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: University of Western Ontario, Canada (Other)
Responsible Party: Principal Investigator, Irina Rachinsky, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R-06-377; 12576 (Registry Identifier: UWO Research Ethics Board number); NCT00972166 (obsolete NCT alias)
Record Dates: First submitted 2008-07-25; First posted 2008-10-16 (Estimated); Last update posted 2012-06-08 (Estimated); Status verified 2012-06

CONDITIONS: Cervical Cancer; Vulvar Cancer
Keywords: Cervical cancer, vulvar cancer, LM/SL, SPECT/CT
MeSH Terms: conditions — Uterine Cervical Neoplasms; Vulvar Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): Single photon emission computed tomography/computed tomography (SPECT/CT) guided lymphatic mapping and sentinel lymphadenectomy (LM/SL) vs. complete lymph node dissection (CLND)
  All cervical cancer and vulvar cancer patients will undergo CLND according to the standard of care in gynecologic cancers as recommended by the International Federation of Gynecology and Obstetrics (FIGO).
  Patients with FIGO IA2 and IB1 cervical cancers will be scheduled for radical hysterectomy and pelvic lymph node dissection.
  Patients with FIGO IB and II vulvar cancers and those of patients with FIGO III with clinically negative regional lymph nodes will be scheduled for vulvectomy and inguinal lymph node dissection.
  Interventions: Device: SPECT/CT guided LM/SL

INTERVENTIONS:
Device: SPECT/CT guided LM/SL — Pre-operatively, SLNs will be detected by low-dose SPECT/CT (99mTc-cystein rhenium colloids, 1cc/1mCi). Intra-operatively, a blue-dye (Patent Blue, 2cc) and a gamma-probe guidance will be used to detect the SLN nodes. All blue-stained and/or hot lymph nodes with a radioactivity greater than 10% of the hottest node will be considered as SLNs. Serial sections of SLNs will be analyzed by H-E staining. In cases of negative H-E, the SLNs will be further analyzed by immunochemistry (CKAE1/CKAE3, and high molecular weight Cytokeratin 34BE12). Non-SLNs will be analyzed as usual in routine by H-E.
  Other Names: Sentinel lymph node detection

SUMMARY:
Nodal staging is a key-step in pre-treatment assessment of gynecological cancers. In recent years, lymphatic mapping and sentinel lymphadenectomy (LM/SL) as a minimally invasive pelvic lymph nodes staging has been successfully evaluated in women with early stage of vulvar cancer, cervical cancer, and endometrial cancer. Such a technique may offer several valuable advantages: a) it is readily applicable in clinical routine using a safe, inexpensive, and reproducible protocol; b) it may help to avoid the cost and the morbidity of unnecessary lymphadenectomy in the majority of cases with uninvolved sentinel lymph nodes; c) it has the potential to guide the surgeon to nodal regions that are not routinely dissected (i.e. pre-sacral, para-aortic nodes) and to identify micro-metastases that would have been ignored otherwise; d) it also offers the basis for sophisticated pathological analysis to detect sub-microscopic nodal metastases using either immunohistochemical or molecular biological techniques.

So far, within the abdomen and the pelvis, the LM/SL technique alone is often blinded to the accurate localization of SLNs. The integration of computed tomography (CT) to single photon emission computed tomography (SPECT) devices in a single gantry (SPECT/CT) has allowed a significant gain in terms of diagnostic accuracy and anatomic precision; clinical examples include malignant melanoma, head and neck cancer, breast cancer, and bladder cancer. In a seminal series of 26 patients with cervical cancer (Zhang et al., 2006), SPECT/CT was recently found superior to conventional planar imaging for detection of SLN and accurate localization. A more recent study (Kushner al., 2007) has also highlighted the technical feasibility and the clinical added-value of a low-dose SPECT/CT in a series of 20 patients with early stage cervical cancer (IA2-IIA) who underwent LM/SL.

In the light of the encouraging data from literature and our own preliminary clinical experience, we hypothesized that the use of LM/SL plus SPECT/CT may be of clinical interest in patients with gynecological cancers.

DETAILED DESCRIPTION:
This clinical trial is aimed at assessing the utility of a minimally invasive surgery preoperatively guided by a new nuclear medicine imaging procedure called SPECT/CT. In patients suffering from an early stage of gynecological cancer with no clinical evidence of lymph node involvement, there is theoretically no reason to perform systematically an aggressive lymphadenectomy as demonstrated for other types of lymphophilic cancers such as malignant melanoma, breast cancer, and head and neck cancer.

We plan to follow a well known and safe procedure in Nuclear Medicine called lymphatic mapping and sentinel lymphadenectomy (LM/SL). The patient will be injected by the gynecologist referee in the department of Nuclear Medicine. These injections consist of a radioactive tracer routinely used in Nuclear Medicine, which allows the detection of the first nodes draining the primary tumor. The so-called sentinel lymph node (SLN) may be different from the lymph nodes anatomically predefined. As well demonstrated for other cancers, including those mentioned above, we hypothesized that the histological status of the SLN may accurately reflect the histological status of the entire nodal basin. If this assumption is clinically validated, the minimally invasive procedure may avoid the cost and the morbidity of unnecessary complete lymph node dissections in the majority of patients with uninvolved SLNs.

The originality of this clinical trial also relies upon the use of a new hybrid imaging device called SPECT/CT, which allows the ability to obtain in a single study both functional and anatomical information. This is critical to precisely guide the surgeon in his task. No contrast medium will be injected during this study. The radiation exposure remains within the limits accepted worldwide; for instance, the CT dose index (CTDI) will be 3.0 mGy, which is in the order of the yearly natural background radiation exposure (< 2mSv).

In this clinical trial, all patients will be treated according to the standard of care currently applied for gynecological cancers. Therefore, either the hysterectomy or the vulvectomy will be followed by a complete lymph node dissection (CLND).

Overall, the research protocol will be carried out in a 1-day protocol including the SPECT/CT guided LM/SL and the CLND.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven gynecological cancers
* Patients with FIGO IA2 and IB1 cervical cancers
* Cervical cancer patients will be scheduled for radical hysterectomy and pelvic lymph node dissection
* Patients with FIGO IB and II vulvar cancers and those of patients with FIGO III with clinically negative regional lymph nodes
* Vulvar cancer patients will be scheduled for vulvectomy and inguinal lymph node dissection
* Informed consent signed by the patient, the gynaecologist, and the nuclear medicine physician referees

Exclusion Criteria:

* Patients with no histological evidence of gynecological cancer
* Patient with regionally advanced disease or metastatic disease
* Patients with clinically and/or radiologically evident regional lymph node metastases
* Patients who are not scheduled for radical surgery and lymph node dissection
* Patients with physical and/or psychological contraindications
* Recent study in Nuclear Medicine with long half-time isotopes (i.e. T ½ >48h; 111In, 67Ga, 201Tl, 131I ) performed within 1 week preceding the LM/SL
* Pregnant or lactating patients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-04; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Sensitivity, predictive value, anatomic localization, and impact on management of SPECT/CT guided LM/SL versus CLND | 6 months -1 year

SECONDARY OUTCOMES:
Patient tolerability and operating time for SPECT/CT guided LM/SL versus CLND | 6 months - 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Irina Rachinsky, MD, MSc, Principal Investigator — The University of Western Ontario - Nuclear Medicine; Jean-Luc Urbain, MD, PhD, Study Chair — The University of Western Ontario - Nuclear Medicine; Monique Bertrand, MD, PhD, Study Director — The University of Western ontario - Gynaecology; Helen Ettler, MD, Study Director — The University of Western Ontario -Pathology
Locations (1):
- 375, South Street Hospital - Dpt. of Nuclear Medicine, London, Ontario, Canada

REFERENCES:
- [Background] Kushner DM, Connor JP, Wilson MA, Hafez GR, Chappell RJ, Stewart SL, Hartenbach EM. Laparoscopic sentinel lymph node mapping for cervix cancer--a detailed evaluation and time analysis. Gynecol Oncol. 2007 Sep;106(3):507-12. doi: 10.1016/j.ygyno.2007.04.031. Epub 2007 Jun 8. PMID 17560635
- [Background] Zhang WJ, Zheng R, Wu LY, Li XG, Li B, Chen SZ. [Clinical application of sentinel lymph node detection to early stage cervical cancer]. Ai Zheng. 2006 Feb;25(2):224-8. Chinese. PMID 16480592
- [Background] Belhocine T, Kridelka F, Thille A, De Barsy C, Foidart-Willems J, Hustinx R, Rigo P. Staging of primary cervical cancers: the role of nuclear medicine. Crit Rev Oncol Hematol. 2003 Jun;46(3):275-84. doi: 10.1016/s1040-8428(03)00027-1. PMID 12791427
- [Background] Van der Zee AG, Oonk MH, De Hullu JA, Ansink AC, Vergote I, Verheijen RH, Maggioni A, Gaarenstroom KN, Baldwin PJ, Van Dorst EB, Van der Velden J, Hermans RH, van der Putten H, Drouin P, Schneider A, Sluiter WJ. Sentinel node dissection is safe in the treatment of early-stage vulvar cancer. J Clin Oncol. 2008 Feb 20;26(6):884-9. doi: 10.1200/JCO.2007.14.0566. PMID 18281661
- [Background] Levenback CF. How safe is sentinel lymph node biopsy in patients with vulvar cancer? J Clin Oncol. 2008 Feb 20;26(6):828-9. doi: 10.1200/JCO.2007.14.7124. No abstract available. PMID 18281651
- [Background] Levenback CF. Status of sentinel lymph nodes in cervical cancer. Gynecol Oncol. 2007 Oct;107(1 Suppl 1):S18-9. doi: 10.1016/j.ygyno.2007.07.039. Epub 2007 Aug 29. No abstract available. PMID 17761270
- [Background] van de Lande J, Torrenga B, Raijmakers PG, Hoekstra OS, van Baal MW, Brolmann HA, Verheijen RH. Sentinel lymph node detection in early stage uterine cervix carcinoma: a systematic review. Gynecol Oncol. 2007 Sep;106(3):604-13. doi: 10.1016/j.ygyno.2007.05.010. Epub 2007 Jul 12. PMID 17628644
- [Background] Benedet JL, Bender H, Jones H 3rd, Ngan HY, Pecorelli S. FIGO staging classifications and clinical practice guidelines in the management of gynecologic cancers. FIGO Committee on Gynecologic Oncology. Int J Gynaecol Obstet. 2000 Aug;70(2):209-62. No abstract available. PMID 11041682
- [Background] Martinez A, Zerdoud S, Mery E, Bouissou E, Ferron G, Querleu D. Hybrid imaging by SPECT/CT for sentinel lymph node detection in patients with cancer of the uterine cervix. Gynecol Oncol. 2010 Dec;119(3):431-5. doi: 10.1016/j.ygyno.2010.08.001. Epub 2010 Sep 6. PMID 20822803
- [Background] Pandit-Taskar N, Gemignani ML, Lyall A, Larson SM, Barakat RR, Abu Rustum NR. Single photon emission computed tomography SPECT-CT improves sentinel node detection and localization in cervical and uterine malignancy. Gynecol Oncol. 2010 Apr;117(1):59-64. doi: 10.1016/j.ygyno.2009.12.021. Epub 2010 Feb 1. PMID 20117827
- [Background] Diaz-Feijoo B, Perez-Benavente MA, Cabrera-Diaz S, Gil-Moreno A, Roca I, Franco-Camps S, Fernandez MS, Garcia-Jimenez A, Xercavins J, Martinez-Palones JM. Change in clinical management of sentinel lymph node location in early stage cervical cancer: the role of SPECT/CT. Gynecol Oncol. 2011 Mar;120(3):353-7. doi: 10.1016/j.ygyno.2010.12.336. Epub 2011 Jan 6. PMID 21215440
- [Background] Freudenberg LS, Gortz E, Hagen C, Harms E, Koska WW, Marlowe RJ, Shadouh S, Stock C. Lymphatic mapping using SPECT/CT in vulvar carcinoma. Clin Nucl Med. 2010 Dec;35(12):950-2. doi: 10.1097/RLU.0b013e3181f9de96. No abstract available. PMID 21206229
- [Background] Kobayashi K, Ramirez PT, Kim EE, Levenback CF, Rohren EM, Frumovitz M, Mar MV, Gayed IW. Sentinel node mapping in vulvovaginal melanoma using SPECT/CT lymphoscintigraphy. Clin Nucl Med. 2009 Dec;34(12):859-61. doi: 10.1097/RLU.0b013e3181becdaf. PMID 20139817
- [Derived] Belhocine TZ, Prefontaine M, Lanvin D, Bertrand M, Rachinsky I, Ettler H, Zabel P, Stitt LW, Sugimoto A, Urbain JL. Added-value of SPECT/CT to lymphatic mapping and sentinel lymphadenectomy in gynaecological cancers. Am J Nucl Med Mol Imaging. 2013;3(2):182-93. Epub 2013 Mar 8. PMID 23526734
- See also: The University of Western Ontario website — http://www.uwo.edu/